CLINICAL TRIAL: NCT02480270
Title: Prospective Clinical and Laboratory Evaluation of Outpatient Antibiotic Treatment for Pulmonary Exacerbations in Children With Cystic Fibrosis
Brief Title: Outpatient Antibiotic Treatment for a Cystic Fibrosis Pulmonary Exacerbation
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0745; UL1TR001082 (NIH)
Record Dates: First submitted 2015-06-15; First posted 2015-06-24 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study plans to learn more about the effect of oral antibiotics for an outpatient pulmonary exacerbation (respiratory illness) on sputum (mucus) bacterial infections, lung function, airway inflammation and quality of life. In this study subjects will perform pulmonary function tests, provide a sputum sample and complete a questionnaire at two separate clinic visits. If a subject is unable to cough up sputum in clinic he or she will be asked to breathe in a salt water solution to help cough up sputum. The first sputum sample will be obtained at the first visit (within 48 hours of starting antibiotics). Pulmonary function testing and the questionnaire will also be completed at this time. Subjects will complete a two week course of oral antibiotics at home. During these two weeks subjects will be asked to write down the times antibiotics are taken and airway clearance (vest treatment) is performed. Within one week of completing the antibiotic course subjects will return to clinic for a second visit. At that time a sputum sample will be obtained again and if subjects are unable to cough up sputum they will again be asked to breathe in salt water solution to help cough up sputum. Pulmonary function testing and the questionnaire will also be completed at this second visit. Sputum samples will be tested for infections with bacteria and viruses. Sputum samples will also be used to measure markers of airway inflammation (swelling). The investigators hypothesize that the use of two weeks of oral antibiotics for the treatment of a pulmonary exacerbation will result in a decrease in the amount of bacteria measured in sputum. Additionally the investigators hypothesize that treatment with antibiotics will lead to an improvement in lung function, a decrease in airway inflammation and an improvement in quality of life measurements.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis based on sweat chloride (≥60) or two known disease causing mutations.
* Age 8 - 18 years
* Starting treatment for an outpatient pulmonary exacerbation
* Willing to participate in study after informed consent and assent has been obtained.

Exclusion Criteria:

* Forced expiratory volume in 1 second (FEV1) less than 40%
* Patients receiving chronic daily oral antibiotics. Patients receiving azithromycin therapy three times a week will not be excluded as its use in this setting is felt to be anti-inflammatory.
* Previous reaction to inhalation of hypertonic saline. This is distinctly unusual in cystic fibrosis.
* Patients who have been treated with oral antibiotics on an outpatient basis within 2 weeks of the exacerbation.
* Patients who are being started simultaneously on inhaled and oral antibiotics. Patients who are routinely receiving inhaled antibiotics as part of their chronic management and continue inhaled antibiotics as previously scheduled will not be excluded.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 30 patients with cystic fibrosis will be recruited from the University of Colorado and Children's Hospital Colorado pediatric cystic fibrosis clinic.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Reduction in bacterial colony count in the primary cystic fibrosis (CF) pathogen identified on culture | Baseline and 3 weeks
  Quantitative measurements of the primary CF pathogen will be obtained on sputum culture at visits 1 and 2. The change in colony count (measured on the log scale) will be used as the primary outcome.

SECONDARY OUTCOMES:
Lung function | Baseline and 3 weeks
  * Change in FEV1 (forced expiratory volume in 1 second).
  * Percent of patients who return to baseline lung function at the completion of an oral antibiotic course (defined as an FEV1 of 95% of baseline or greater).
Airway inflammation | Baseline and 3 weeks
  Change in measurements of sputum total white blood cell count, neutrophil count, neutrophil elastase, LTB4 (leukotriene B4), IL-8 (interleukin 8), IL-1B (interleukin 1, beta)
Quality of Life | Baseline and 3 weeks
  Change in patient reported symptoms and severity (Cystic Fibrosis Questionnaire-Revised)
Microbiome | Baseline and 3 weeks
  Change in airway microbiota in sputum samples obtained before and after oral antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Jordana E Hoppe, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States